CLINICAL TRIAL: NCT01524848
Title: Pazopanib in Advanced GISTs Refractory to Imatinib and Sunitinib - A Non-comparative Phase II Multicenter Study by the Scandinavian Sarcoma Group
Brief Title: Pazopanib in Advanced Gastrointestinal Stromal Tumors Refractory to Imatinib and Sunitinib
Acronym: PAGIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scandinavian Sarcoma Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSG XXI
Record Dates: First submitted 2012-01-24; First posted 2012-02-02 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2016-05

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Clinical trial; Investigational drugs; Gastrointestinal stromal tumors; Pazopanib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label (Other): Single arm pazopanib
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Two (2) tablets of 400 mg given once daily continuously
  Other Names: Votrient

SUMMARY:
Patients with metastatic or locally advanced gastrointestinal stromal tumors (GIST) who develop resistance against the two hitherto approved drugs for this disease, the tyrosin kinase inhibitors (TKIs) imatinib and sunitinib, have a poor prognosis. Sometimes a further response may be achieved by other drugs, mainly other TKIs, which have been explored in different studies but not yet have been approved for clinical use. Pazopanib is a TKI inhibiting the tyrosin kinases KIT, PDGFRA, and VEGF 1-3, all of which have important roles in the pathogenesis of GIST. Theoretically, it may function in GIST, and it deserves investigational trials. The drug is approved for metastatic renal cancer and is relatively well tolerated. In this trial (SSG XXI), the disease control rate (DCR) = (CR+PR+SD) after 12 weeks of treatment will be assessed as the primary endpoint, and at the same time trough levels will be measured. Secondary endpoints include ORR, PFS, toxicity, and disease control rate in relation to trough level week 12 and in relation to the primary mutation of the tumor (if known). The goal is to include 72 patients in the trial, which is open and single arm.

ELIGIBILITY:
Eligibility Criteria:

* Metastatic and/or locally advanced GIST, with diagnosis based on histology with positive c-kit and/or DOG-1, or with a GIST-typical mutation in KIT or PDGFR
* Measurable disease on CT (computed tomography) as defined by RECIST criteria; at least one measurable lesion not given radiotherapy
* History of progressive disease on CT according to RECIST criteria after both imatinib and sunitinib treatment, and also after nilotinib if this drug has been given
* No other TKIs given than imatinib, sunitinib and nilotinib
* Age at least 18 years at the time of diagnosis of GIST
* WHO performance status 0-2
* Resolution of all toxic side effects from earlier TKI treatment and any other potential non-TKI treatment to grade 1 or below
* Sufficient organ functions as defined in the protocol
* Absence of earlier or present certain other conditions as defined in the protocol
* No pregnancy or lactation
* Women with childbearing potential must accept the use of adequate contraception throughout the study period
* Written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-01 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Disease control rate | Week 12
  The ratio of patients with CR (complete remission) + PR (partial remission) + SD (stable disease) at week 12 after start of treatment

SECONDARY OUTCOMES:
Progression free survival (PFS) | The patients will be followed for the duration of the trial treatment, an expected average of 6 months
  Progression free survival (KM analysis) for all patients administered the study drug
DCR in relation to mutation | Week 12
  Disease control rate as described above in relation to the type of mutation of the primary tumor if this is available (not mandatory)
DCR in relation to plasma concentration | Week 12
  Disease control rate as defined above in relation to the trough level (plasma concentration) of the study drug at week 12
Toxicity | The patients will be followed for the duration of the trial treatment + 1 month, an expected average of 7 months
  Recording of adverse events including SAE/SAR for all patients administered the study drug
Overall response rate | The patients will be followed for the duration of the trial treatment, an expected average of 6 months
  ORR = CR+PR at the time of best response during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Eriksson, MD PhD, Principal Investigator — Scandinavian Sarcoma Group
Locations (16):
- Denmark (2):
  - Aarhus University Hospital, dept. of Oncology, Aarhus
  - Herlev Hospital, dept. of Oncology, Herlev
- Finland (2):
  - Helsinki University Hospital, dept. of oncology, Helsingfors
  - Kuopio University Hospital Cancer Center, Kuopio
- Germany (3):
  - Klinik für Interdisziplinäre Onkologie, Sarkomzentrum Berlin-Brandenburg, Berlin
  - Universitätsklinikum Essen, Innere klinik und Poliklinik, Essen
  - Studienzentrale chirurgische klinik, Universitäts medizin Mannheim, Mannheim
- Norway (3):
  - Dept of Oncology, Haukeland University Hospital, Bergen
  - Norwegian Radium Hospital, Oslo
  - Dept of Oncology, St Olav Hospital, Trondheim
- Sweden (6):
  - Dept of Oncology, Sahlgrenska University Hospital, Gothenburg
  - Dept of Oncology, Linköping University Hospital, Linköping
  - Dept of Oncology, Skane University Hospital, Lund
  - Radiumhemmet, Karolinska University Hospital, Stockholm
  - Dept of Oncology, Norrland University Hospital, Umeå
  - Dept of Oncology, Academic Hospital, Uppsala